CLINICAL TRIAL: NCT05201170
Title: A Phase 3, Multi-center, Randomized, Double-Masked and Vehicle-Controlled Study Evaluating the Efficacy and Safety of the Melanocortin, PL9643 Ophthalmic Solution, Compared to Vehicle in Subjects with Dry Eye
Brief Title: A Phase 3, Multi-Center Study Evaluating PL9643 in Patients with Dry Eye
Acronym: MELODY-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Palatin Technologies, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PL9643-301
Record Dates: First submitted 2022-01-08; First posted 2022-01-21 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2022-01

CONDITIONS: Dry Eye; Dry Eye Syndromes
Keywords: Dry eye; Ophthalmology; Eye diseases; Corneal diseases; Conjunctival diseases; Ophthalmic Solutions; Pharmaceutical Solutions
MeSH Terms: conditions — Dry Eye Syndromes; Eye Diseases; Corneal Diseases; Conjunctival Diseases

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to either the PL9643 treatment group or to the vehicle control group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All individuals involved in the conduct of the study, and the enrolled patients, will remain masked to the randomized study treatment assignments until the database is unmasked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PL9643 Ophthalmic Solution (Experimental): PL9643 ophthalmic solution bilaterally three times a day.
  Interventions: Drug: PL9643 Ophthalmic Solution
- Vehicle Ophthalmic Solution (Active Comparator): Vehicle ophthalmic solution bilaterally three times a day.
  Interventions: Drug: Vehicle Ophthalmic Solution

INTERVENTIONS:
Drug: Vehicle Ophthalmic Solution — Ophthalmic Solution
  Other Names: Control
  Arms: Vehicle Ophthalmic Solution
Drug: PL9643 Ophthalmic Solution — Ophthalmic Solution
  Other Names: Active study medication
  Arms: PL9643 Ophthalmic Solution

SUMMARY:
This is a multi-center, double-masked, randomized, vehicle-controlled study testing PL9643, an ophthalmic solution to determine if safe and efficacious for dry eye patients.

After a 2-week run-in period, patients will be randomized equally to the PL9643 ophthalmic solution or vehicle ophthalmic solution administered bilaterally three times a day for 12 weeks.

A Data Monitoring Committee was engaged to review interim data.

DETAILED DESCRIPTION:
This is a multi-center, double-masked, randomized, vehicle-controlled study testing PL9643, an ophthalmic solution, to determine the safety and efficacy against a vehicle in dry eye patients.

During a 2-week/14-day study run-in period (for the purpose of subject selection) prior to randomization, all subjects will receive Vehicle Ophthalmic Solution (vehicle) bilaterally three times a day. Randomization will then occur in a 1:1 ratio where patients will be assigned to receive PL9643 ophthalmic solution given bilaterally three times a day or vehicle ophthalmic solution administered bilaterally three times a day. The treatment period is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age;
2. Provide written informed consent;
3. Be willing and able to comply with all study procedures;
4. Have a patient-reported history of dry eye for at least 5 years prior to Visit 1;
5. Have a history of use or desire to use eye drops for dry eye symptoms within 6 months of Visit 1;
6. Have a best corrected visual acuity (BCVA) of 0.7 logarithm of the minimum angle of resolution (logMAR) or better (Snellen equivalent score of 20/100 or better) in each eye at Visit 1;
7. Have an inferior fluorescein corneal staining score > 1 at both Visits 1 and 2 Pre-CAE®;
8. Have an Eye Discomfort from the Visual Analog Scale (VAS) ≥25 at both Visits 1 and 2 Pre-CAE®;
9. Report a score of ≥ 2 according to the Ora Calibra® Ocular Discomfort & 4-Symptom Questionnaire in at least one of the dry eye symptoms at Visits 1 and 2 Pre-CAE®;
10. Have a Schirmer's Test score of ≤ 10 mm and ≥ 1 mm at Visits 1 and 2;
11. Have a corneal fluorescein staining score of ≥ 2 in any corneal region (inferior, central or superior) according to the Ora Calibra® Corneal and Conjunctival Staining Scale for Grading of Fluorescein Staining in at least one eye at Visits 1 and 2 Pre-CAE®;
12. Have a conjunctival redness score ≥ 1 according to the Ora Calibra® Conjunctival Redness for Dry Eye Scale in at least one eye at Visits 1 and 2 Pre-CAE®;
13. Demonstrate in the same eye(s) a response to the CAE®at Visits 1 and 2 as defined by:

    1. Having at least a ≥1 point increase in fluorescein staining in the inferior region in at least one eye following CAE® exposure;
    2. Reporting an Ocular Discomfort score ≥3 at 2 or more consecutive time points in at least one eye during CAE® exposure (if a subject has an Ocular Discomfort rating of 3 at time = 0 for an eye, s/he must report an Ocular Discomfort rating of 4 for two consecutive measurements for that eye). Note: a subject cannot have an Ocular Discomfort score of 4 at time = 0);
14. Have at least one eye, the same eye, satisfy all criteria for 7, 8, 9, 10, 11, 12 and 13 above;
15. A negative urine pregnancy test if female of childbearing potential (those who are not surgically sterilized [bilateral tubal ligation, hysterectomy or bilateral oophorectomy] or post-menopausal [12 months after last menses]) and must use adequate birth control through the study period. For non-sexually active females, abstinence may be regarded as an adequate method of birth control

Exclusion Criteria:

1. Have any clinically significant slit-lamp findings at Visit 1 that may include active blepharitis, meibomian gland dysfunction, lid margin inflammation, or active ocular allergies that require therapeutic treatment, and/or in the opinion of the Investigator may interfere with study parameters;
2. Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation at Visit 1 or Visit 2;
3. Have worn contact lenses within 7 days of Visit 1 or anticipate using contact lenses during the study;
4. Have previously had laser-assisted in situ keratomileusis (LASIK) surgery within the last 12 months;
5. Have used Restasis®, Xiidra®, Cequa®, or Eysuvis® within 60 days of Visit 1;
6. Have had any ocular and/or lid surgeries in the past 6 months or have any planned ocular and/or lid surgeries over the study period;
7. Have had any laser procedures (e.g. YAG capsulotomy) in the past 3 months;
8. Be using or anticipate using temporary punctal plugs during the study that have not been stable within 30 days of Visit 1;
9. Be currently taking any topical ophthalmic prescription (including medications for glaucoma) or over-the-counter solutions, artificial tears, gels or scrubs, and cannot discontinue these medications for the duration of the trial (excluding medications allowed for the conduct of the study); the respective wash-out periods are required for thefollowing medications:

   1. Ocular, oral or nasal antihistamines: 72 hours prior to Visit 1 and during the study.
   2. Oral aspirin or aspirin-containing products allowed if dose has been stable over past 30 days prior to Visit 1 and no change in dose is anticipated during the study period
   3. Corticosteroids or mast cell stabilizers (including ocular): 14 days prior to Visit 1
   4. Any medication (oral or topical) known to cause ocular drying that has not been administered as a stable dose for at least 30 days prior to Visit 1 and during the study
   5. All other topical ophthalmic preparations (including artificial tear substitutes) other than the study drops: 72 hours prior to Visit 1
10. Have an uncontrolled systemic disease;
11. Be a woman who is pregnant, nursing, or planning a pregnancy;
12. Be unwilling to submit a urine pregnancy test at Visit 1 and Visit 6 (or early termination visit) if of childbearing potential. Non-childbearing potential is defined as a woman who is permanently sterilized (e.g., bilateral tubal ligation, hysterectomy or bilateral oophorectomy), or is post-menopausal (without menses for 12 consecutive months);
13. Be a woman of childbearing potential who is not using an acceptable means of birth control; acceptable methods of contraception include: hormonal - oral, implantable, injectable, or transdermal contraceptives; mechanical - spermicide in conjunction with a barrier such as a diaphragm or condom; intrauterine device; or surgical sterilization of partner. For non-sexually active females, abstinence may be regarded as an adequate method of birth control; however, if the subject becomes sexually active during the study, she must agree to use adequate birth control as defined above for the remainder of the study;
14. Have a known allergy and/or sensitivity to the test article or its components;
15. Have a condition or be in a situation which the Investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study;
16. Have used an investigational drug or device within 30 days of Visit 1 unless the Investigator or Sponsor deems a washout period of up to 60 days is required;
17. Participated in a previous clinical study involving PL9643;
18. Be unable or unwilling to follow instructions, including participation in all study assessments and visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 575 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-11-21 (Actual)

PRIMARY OUTCOMES:
Conjunctival Sum Lissamine Green Staining | Visit 6 (Day 85), Change from Pre-CAE to Post-CAE
  Measured by the Ora Calibra® Scale. Change from Baseline to week 12.
Ocular Pain | Change from Pre-CAE to Post-CAE at Visit 6 (Day 85)
  As Measured by Visual Analog Scale (VAS). PL9643 versus Vehicle, in hyper-responder sub-population. Hyper-responder sub-population is defined as those patients achieving a VAS score of 4 or greater within the first 30 minutes of being challenged in the CAE® (clinical symptom) at Visit 2.

SECONDARY OUTCOMES:
Nasal Lissamine Green Staining in Study Eye | Change from Baseline to Visit 6 (Day 85), Pre-CAE
  As measured by Ora Calibra Scale at Visit 6 (Day 85) in Study Eye
Tear Film Break-Up Time (TFBUT) in Study Eye | Change from Baseline to Visit 6 (Day 85), Post-CAE
  Change from Baseline Post-CAE® to Week 12 Post-CAE®
Total Sum Lissamine Green Staining in Study Eye | Change from Baseline Pre-CAE® to Week 12 Pre-CAE
  As measured by Ora Calibra Scale at Visit 6 (Day 85) in Study Eye
Ocular Pain for ITT | Visit 6 (Day 85), Change from Pre-CAE to Post-CAE
  As Measured by Visual Analog Scale at Visit 6 (Day 85), PL9643 versus Vehicle, In ITT population
Inferior Fluorescein Staining in Study Eye | Change from Baseline to Visit 6 (Day 85), Post-CAE
  As Measured by Ora Calibra Scale at Visit 6 (Day 85) in Study Eye
Inferior Corneal Fluorescein Staining in Study Eye | Change from Baseline to Visit 6 (Day 85), Pre-CAE
  As measured by Ora Calibra Scale at Visit 6 (Day 85) in Study Eye
Foreign Body Sensation for Hyper-Responders | Visit 6 (Day 85), Change from Pre-CAE to Post-CAE
  As Measured by Visual Analog Scale at Visit 6 (Day 85) for Hyper-Responders
Eye Dryness for Hyper-Responders versus Vehicle in hyper-responder sub-population | Change from Baseline to Visit 6 (Day 85), Post-CAE
  As Measured by Visual Analog Scale at Visit 6 (Day 85) for Hyper-Responders
Unanesthetized Schirmer Test Result (mm) in Study Eye | Change from Baseline to Visit 6 (Day 85), Pre-CAE
  Measured at Visit 6 (Day 85) in Study Eye
Eye Discomfort for Hyper-responders versus Vehicle in hyper-responder sub-population | Change from Baseline to Visit 6 (Day 85), Post-CAE
  As Measured by Visual Analog Scale at Visit 6 (Day 85) for Hyper-responders

OTHER OUTCOMES:
Pain for Hyper-Responders | Change from Baseline to Visit 3 (Day 15), Post-CAE
  As Measured by Visual Analog Scale at Visit 3 (Day 15) for Hyper-Responders
Pain for ITT | Visit 3 (Day 15), Change from Pre-CAE to Post-CAE
  As Measured by Visual Analog Scale at Visit 3 (Day 15) PL9643 versus Vehicle, In ITT population
Eye Discomfort for Hyper-responders | Visit 3 (Day 15), Change from Pre-CAE to Post-CAE
  As Measured by Visual Analog Scale, Pre-CAE at Visit 3 (Day 15) for Hyper-responders

CONTACTS AND LOCATIONS:
Overall Officials: Brian Dodge, Study Director — Palatin
Locations (18):
- United States (18):
  - Global Research Management, Glendale, California
  - Eye Research Foundation, Newport Beach, California
  - East West Eye Institute, Torrance, California
  - Pankratz Eye Institute, Columbus, Indiana
  - Michael Washburn Center for Ophthalmic Research, LLC, Indianapolis, Indiana
  - Kentucky Eye Institute, Lexington, Kentucky
  - Butchertown Clinical Trials, Louisville, Kentucky
  - Andover Eye Associates, Andover, Massachusetts
  - Center for Sight, Las Vegas, Nevada
  - Mint Hill, Mint Hill, North Carolina
  - Core, Inc, Shelby, North Carolina
  - Bergstrom Eye research, LLC, Fargo, North Dakota
  - Erie Retina Research, LLC, Erie, Pennsylvania
  - Advancing Vision Research, Goodlettsville, Tennessee
  - Total Eye Care, PA, Memphis, Tennessee
  - Advancing Vision Research, Smyrna, Tennessee
  - Austin Clinical Research, Austin, Texas
  - Axis Clinical, Dallas, Texas